CLINICAL TRIAL: NCT00268177
Title: A 13-week, Double-blind, Parallel Group, Multi-centre Study to Compare the Bronchial Anti-inflammatory Activity of the Combination of Salmeterol/Fluticasone Propionate 50/500mcg Twice Daily Compared With Placebo Twice Daily in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Airway Inflammation In Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO30005
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Airways; Pulmonary; Obstructive; Chronic; inflammation; salmeterol/fluticasone propionate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Inflammation | interventions — Salmeterol Xinafoate; Fluticasone

INTERVENTIONS:
Drug: Salmeterol/fluticasone propionate 50/500mcg Diskus

SUMMARY:
This study was designed to look at effects of salmeterol/fluticasone propionate compared to placebo on airway inflammation in patients with chronic obstructive airways disease

ELIGIBILITY:
Inclusion Criteria:

* Established clinical history of chronic obstructive airways disease.
* Must be current or ex-smokers with a smoking history of at least 10 pack-years (e.g. 20 cigarettes/day for 10 years or 10 cigarettes/day for 20 years).
* Must have reduced lung function, defined as a Forced Expiratory Volume in 1 second (FEV1) of between 40-80% of predicted normal values.

Exclusion Criteria:

* Diagnosis of any other serious disease and must have a chest X-ray to eliminate a diagnosis other than COPD.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2002-10; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
To compare the number of CD68+ and CD8+ inflammatory cells per area of biopsy tissue and the percentage and total number of neutrophils in induced sputum between salmeterol/fluticasone propionate and placebo

SECONDARY OUTCOMES:
To compare the number of mast cells, CD45+,CD4+,IFN-gamma mRNA+,TNF-alpha mRNA+, per area of biopsy and the percentage and number of macrophages, eosinophils, lymphocytes in induced sputum between salmeterol/fluticasone propionate and placebo

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Denmark (2):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, København NV
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- GSK Investigational Site, Helsinki, Finland
- GSK Investigational Site, Palermo, Sicily, Italy
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
- Spain (2):
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Madrid
- United Kingdom (5):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Norwich, Norfolk
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Hull
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Barnes NC, Qiu Y, Zhu J, et al. Anti-inflammatory effects of salmeterol/fluticasone propionate (SFC) by smoking status in COPD. Eur Respir J 2005; 26(suppl 49): 204S.
- [Background] Barnes NC, Qiu YS, Pavord I. Clinical improvement with salmeterol/fluticasone proprionate is associated with reduction in inflammation in patients with COPD. European Respiratory Journal Supplement 2005; 26(Suppl. 49): 717 (plus poster) Abstract P4574.
- [Background] Barnes NC, Qiu YS, Pavord ID, Parker D, Davis PA, Zhu J, Johnson M, Thomson NC, Jeffery PK; SCO30005 Study Group. Antiinflammatory effects of salmeterol/fluticasone propionate in chronic obstructive lung disease. Am J Respir Crit Care Med. 2006 Apr 1;173(7):736-43. doi: 10.1164/rccm.200508-1321OC. Epub 2006 Jan 19. PMID 16424444
- [Background] Baseline characteristics of the first 5,000 copd patients enrolled in the torch survival study. Calverley, P. M. A., Celli, B., Ferguson, G., Jenkins, C., Jones, P., Pride, N. B., Vestbo, J., Anderson, J., and Pauwels, R. 13th Annual Congress of the European Respiratory Society 9/27/2003 Vienna; Austria
- [Background] Pavord I, Parker D, Barnes NC, et al. Effects of salmeterol/fluticasone propionate (SFC) on airway inflammation in induced sputum in COPD. Eur Respir J 2005; 26(suppl 49): 203S.
- [Background] Qiu Y, Davis P, Zhu J, et al. Anti-inflammatory effects of salmeterol/fluticasone propionate (SFC) on airway T-lymphocyte populations in COPD. Eur Respir J 2005; 26(suppl 49): 203S.
- [Background] Qiu Y, Davis P, Zhu J, et al. Effects of salmeterol/fluticasone propionate (SFC) on airway inflammation in COPD: a placebo-controlled study of endobronchial biopsies. Eur Respir J 2005; 26(suppl 49): 203S.
- [Background] Vestbo J; TORCH Study Group. The TORCH (towards a revolution in COPD health) survival study protocol. Eur Respir J. 2004 Aug;24(2):206-10. doi: 10.1183/09031936.04.00120603. PMID 15332386
- [Background] Zhu J, Qiu Y, Barnes NC, Johnson M, Pavord I, Jeffery P. The effect of salmeterol/fluticasone propionate (SFC) on pro-inflammatory gene expression in COPD. PATS 2005; 2(abstracts issue): A127
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: SCO30005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SCO30005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCO30005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCO30005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCO30005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SCO30005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCO30005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register